CLINICAL TRIAL: NCT02792881
Title: The Safety, Feasibility and Oncological Outcomes of Laparoscopic Completion Total Gastrectomy for Remnant Gastric Cancer: A Prospective Trial (FUGES-004)
Brief Title: The Safety, Feasibility and Oncological Outcomes of Laparoscopic Completion Total Gastrectomy for Remnant Gastric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Professor, Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FUGES-004
Record Dates: First submitted 2016-05-26; First posted 2016-06-08 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Remnant Gastric Cancer
Keywords: Laparoscopic Completion Total Gastrectomy; Remnant gastric cancer; Feasibility; Prognosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laparoscopic Completion Total Gastrectomy Group (Experimental): Patients who underwent laparoscopic completion total gastrectomy with D2 lymphadenectomy will be assigned to this group.
  Interventions: Procedure: Laparoscopic completion total gastrectomy with D2 lymphadenectomy

INTERVENTIONS:
Procedure: Laparoscopic completion total gastrectomy with D2 lymphadenectomy — After exclusion of T4b, bulky lymph nodes, or distant metastasis case by diagnostic laparoscopy, Laparoscopic completion total gastrectomy with D2 lymphadenectomy will be performed with curative treated intent. For carcinomas arising in the remnant stomach with a gastrojejunostomy, jejunal lymph nodes adjacent to the anastomosis are included as regional lymph nodes. The type of reconstruction will be selected according to the surgeon's experience and the anastomotic procedure will be performed extracorporeally through an auxiliary incision.

SUMMARY:
This study aims to investigate the safety, feasibility, and long-term oncological outcomes of laparoscopic completion total gastrectomy for remnant gastric cancer.

DETAILED DESCRIPTION:
In 2005, since Yamada reported the first case of laparoscopic completion total gastrectomy (LCTG) for RGC, laparoscopic technology was widely used in the treatment of RGC. However, due to the low incidence and rapid aggravation of RGC, adhesion, anatomic changes, and more complex lymphatic pathways caused by the previous operation, the popularity of LCTG is limited. Therefore, higher level evidence is warranted to further confirm the safety, feasibility, and oncological outcomes of LCTG in patients with RGC. This prospective single-arm study is designed to evaluate the safety, feasibility, and long-term oncological outcomes of laparoscopic completion total gastrectomy for remnant gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

Age between 18 and 75 years; Carcinomas arise in the remnant stomach following gastrectomy, irrespective of the histology of the primary lesion (benign or malignant) or its risk of recurrence, the extent of resection, or the method of reconstruction; cT1-4a, N-/+, M0 at preoperative evaluation according to the AJCC Cancer Staging Manual, 7th Edition; Performance status of 0 or 1 on ECOG scale; ASA class I, II, or III; Written informed consent.

Exclusion Criteria:

Distant metastasis in the preoperative examinations; Previous upper abdominal surgery (except laparoscopic cholecystectomy, previous gastrectomy, endoscopic mucosal resection or endoscopic submucosal dissection); Other malignant diseases (except gastric cancer) within the past 5 years; Enlarged or bulky regional lymph node (diameter over 3cm) supported by preoperative imaging including enlarged or bulky No.10 lymph nodes; Women during breast-feeding or pregnancy; Severe mental disorder; Unstable myocardial infarction, angina, or cerebrovascular accident within the past 6 months; History of continuous systematic administration of corticosteroids within one month; FEV1<50% of predicted values; Requirement of simultaneous surgery for other disease; Emergency surgery due to complications (bleeding, obstruction, or perforation) caused by gastric cancer.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Morbidity | 30 days
  The early postoperative complication are defined as the event observed within 30 days after surgery.

SECONDARY OUTCOMES:
3-year disease free survival rate | 36 months
3-year overall survival rate | 36 months
3-year recurrence pattern | 36 months
  Recurrence patterns are classified into five categories at the time of first diagnosis: locoregional, hematogenous, peritoneal, distant lymph node, and mixed type
Mortality | 30days
  The early mortality are defined as the event observed within 30 days after surgery.
Rates of combined organ resection | 1 day
  Combined organ resection performing by severe injury or abdominal adhesions
Intraoperative morbidity rates | 1 day
  With the number of patients undergoing surgery as the denominator, the number of patients with any of the following intraoperative complications is calculated as numerator.
Number of retrieved lymph nodes | 1 day
  Number of retrieved lymph nodes
Operation time | 1 day
  From skin incision to skin closure
Postoperative recovery course | 10 days
  Including time to first flatus, time to initiation of solid food intake, time to removal of intra-abdominal drains, hospital stay
Intraoperative blood loss | 1 day
Inflammatory and immune response and nutrional status | 7 days
  the values of hemoglobin, prealbumin, albumin, C-reactive protein, and white blood cell count from peripheral blood before the operation and on postoperative day 1, 3, 5 are recorded.
Textbook Outcome | 30 days
  Textbook outcome (TO) was defined based on review of existing TO metrics in the literature including outcomes such as complete-potentially curative status, no intraoperative complications, no eventful postoperative complications (Clavien-Dindo grade III or higher), 15 lymph nodes(LNs) examined, hospital stay < 21days, no reintervention (surgical, endoscopic or radiological) within 30 days after surgery, no readmission to the intensive care unit (ICU) within 30 days after surgery, no postoperative mortality within 30 days after surgery, and no hospital readmission within 30 days after discharge. When all nine desired health outcomes were realized, TO was achieved.
Technical performance | 1 day
  Technical performance were assessed by the Objective Structured Assessments of Technical Skills (OSATS) and the Generic Error Rating Tool.
The Surgery Task Load Index (SURG-TLX) | 1 day
  Surgeons were required to complete one modified SURG-TLX questionnaire for each procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Changming Huang, M.D.,Ph.D., Study Chair — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

REFERENCES:
- [Derived] Wu D, Zhong Q, Zhang ZQ, Liu SQ, Qiu TY, Chen JY, Jiang YM, Lin GT, Liu ZY, Shang-Guan ZX, Sun YQ, Zheng CH, Li P, Xie JW, Lin JX, Chen QY, Huang CM. Comprehensive comparison of technical performance, surgical outcomes, and oncologic prognosis between remnant gastric cancer and primary upper-third gastric cancer in the era of minimally invasive surgery: A pooled analysis of 3 prospective trials. Surgery. 2025 Jul;183:109395. doi: 10.1016/j.surg.2025.109395. Epub 2025 May 8. PMID 40344992
- [Derived] Zhong Q, Wu D, Jiang YM, He QL, Dang XY, Xu DB, Sun YQ, Su GQ, Guo KQ, Cai LS, Zhang HX, Ye W, Lin GT, Li P, Xie JW, Chen QY, Zheng CH, Lu J, Huang CM, Lin JX. The safety, feasibility, and oncological outcomes of laparoscopic completion total gastrectomy for remnant gastric cancer: a prospective study with 3-year follow-up (FUGES-004 study). Int J Surg. 2024 Jun 1;110(6):3382-3391. doi: 10.1097/JS9.0000000000001388. PMID 38597388